CLINICAL TRIAL: NCT06849765
Title: Feasibility and Safety Validation Study of a Rehabilitation Program and Platform Using Digital Devices for Recovery of Bedridden Patients
Brief Title: Feasibility and Safety of Digital Rehab Platform for Bedridden Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: EverEx Inc. (Industry)
Responsible Party: Principal Investigator, Won Kim, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2024-1729-0002
Record Dates: First submitted 2024-12-02; First posted 2025-02-27 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: ICU Acquired Weakness (ICUAW)
Keywords: Intensive Care Unit Acquired weakness; Digital Therapeutics
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): The rehabilitation program will utilize the MORA app to create individualized interventions based on each patient's physical capabilities.
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation — The rehabilitation program will utilize the MORA app to create individualized interventions based on each patient's physical capabilities.

SUMMARY:
Study Title Rehabilitation Program for Bedridden Patients Using Digital Devices

Study Purpose This study aims to evaluate the effectiveness of a rehabilitation program using digital devices and apps for bedridden patients in a hospital setting. The goal is to determine if digital rehabilitation can help improve physical function and contribute to recovery for patients who are unable to move easily.

Study Participants The study will involve 20 adult patients who are bedridden and hospitalized. Participants will use the provided app, which delivers a customized rehabilitation exercise program.

Study Methodology Exercise Protocol: Patients will follow a personalized exercise program through the MORA app, performing the exercises twice daily for a period of 2 weeks. Each session will last approximately 30 minutes and will be tailored to the patient's physical condition to ensure safety.

Safety and Effectiveness Monitoring: The study will track the patients' physical function (e.g., strength, mobility) and monitor for any discomfort or adverse effects that may arise during the exercise sessions.

Study Duration The study will run from September 2024 to December 2025. During this period, participants will engage in rehabilitation exercises using the digital app.

Expected Outcomes This study will demonstrate whether digital rehabilitation can be a safe and effective treatment option for bedridden patients in the hospital. The findings are expected to help improve physical recovery for these patients and contribute to enhancing rehabilitation practices within hospital settings.

Safety Considerations The exercises in this study are designed with safety in mind and will be adjusted to a low intensity. Any discomfort or adverse effects will be monitored closely, and immediate action will be taken if necessary. All exercises will be conducted under the supervision of healthcare professionals.

DETAILED DESCRIPTION:
Summary of the Research Plan Title: Feasibility and Safety Validation Study of a Rehabilitation Program and Platform Using Digital Devices for Recovery of Bedridden Patients

Objectives:

This study aims to analyze the physical function characteristics of bedridden patients and to develop a rehabilitation program using the MORA app to validate the feasibility and safety of the rehabilitation program and platform.

Principal Investigator: Dr. Kim Won Co-investigators: Dr. Cha Seungwoo, Dr. Lee Chaerin Institution: Seoul Asan Medical Center Study Participants: Hospitalized patients at Seoul Asan Medical Center with a Functional Ambulatory Category (FAC) score of 3 or below and bedridden.

Study Design: A prospective cohort clinical study involving 20 participants who meet the inclusion and exclusion criteria.

Evaluation Method: The rehabilitation program will be customized based on each patient's condition using the MORA app. The intervention will last for two weeks, with two sessions per day (morning and afternoon), each lasting up to 30 minutes. For the first five days, researchers will directly visit participants to monitor app usage and physical movements. Afterward, participants will continue independently with reminders via push notifications, phone calls, or visits. Pre-intervention, 1-week, and 2-week assessments will be conducted to evaluate various parameters.

1. Research Background Many hospitalized patients become bedridden after surgery, resulting in muscle weakness and complications such as pneumonia (Herridge, Margaret S., et al., 2011). Prolonged immobility can lead to decreased mobility, shortened life expectancy, and increased risk of long-term care admission (Guralnik JM, et al., 2011). Although hospitals offer rehabilitation treatments for bedridden patients, there are significant challenges due to limited resources and low insurance reimbursements. As a result, many bedridden patients do not receive adequate rehabilitation care.

   While there are some rehabilitation devices available for bedridden patients, they are often costly and require professional staff for operation, limiting their accessibility. In light of these challenges, there is a need for accessible, self-guided rehabilitation approaches that encourage active movement. Mobile platforms utilizing digital rehabilitation technologies have emerged as a promising solution to overcome these limitations. In the U.S., digital therapies have been shown to reduce pain and improve symptoms of depression and anxiety in patients with back pain (Shebib et al., 2019). However, digital rehabilitation platforms for bedridden patients are still lacking.

   Digital rehabilitation platforms can help overcome the spatial and economic limitations of face-to-face therapy and are a promising solution to the rehabilitation program shortage for bedridden patients. These platforms also provide an opportunity for easy monitoring, data collection, and physical function assessment. Therefore, the purpose of this study is to validate the feasibility and safety of a digital rehabilitation program and platform for bedridden patients.
2. Research Objectives To develop a rehabilitation program and platform for bedridden patients and validate its feasibility and safety.
3. Expected Study Duration The study is expected to be conducted from the date of IRB approval through December 31, 2025.
4. Study Participants and Methods 1) Study Participants

Inclusion Criteria:

Adults aged 19 years or older hospitalized at Seoul Asan Medical Center Bedridden patients with a FAC score of 3 or below (patients who need assistance from a caregiver for walking without physical contact).

Exclusion Criteria:

Patients unable to operate the app due to cognitive impairment Patients experiencing significant pain or limitations in range of motion Biomechanically unstable patients Patients with severe visual or auditory impairments that prevent participation in rehabilitation exercises.

Target Sample Size and Rationale:

This study is a pilot study, and based on similar past studies, the expected sample size is 20 participants, considering the study duration and available participants at Seoul Asan Medical Center.

2) Research Methods The study will recruit patients who meet the inclusion and exclusion criteria. A personalized rehabilitation program will be developed using the MORA app. The intervention will last for two weeks, with two sessions per day (morning and afternoon), each lasting no longer than 30 minutes. During the first five days, the research team will visit participants to monitor the app's functionality and physical exercises. Afterward, participants will be reminded to perform exercises independently via push notifications, phone calls, or visits. The research team will assess various parameters before, one week after, and two weeks after the intervention.

5. Statistical Analysis Principles and Methods Statistical analysis will be conducted using SPSS and R software with a significance level set at p < 0.05. Descriptive statistics will summarize patient characteristics and physical function. For categorical variables, chi-square tests and logistic regression will be used, while continuous variables will be analyzed using Mann-Whitney U tests, Kruskal-Wallis tests, and Spearman correlation.

6. Participant Withdrawal Criteria

Participants may withdraw from the study at any time. Other criteria for withdrawal include:

Participant or legal guardian requests withdrawal Discovery that the participant is no longer eligible or suitable for the study Determination by the investigator or ethics committee that continuation is inappropriate.

7. Expected Adverse Effects Possible adverse effects include temporary breathlessness, tachycardia, blood pressure changes, falls, and device dislodgement. However, since the intervention involves low-intensity exercises, the likelihood of serious adverse effects is low. The risk of falls is considered minimal compared to rehabilitation performed outside the bed.

8. Early Termination Criteria

The study may be terminated early under the following conditions:

Participant withdrawal Discovery that the participant is unsuitable for the study Investigator or ethics committee judgment that the study should be discontinued If the ethics committee or institution decides the trial should be halted. 9. Ethical Considerations This study will be conducted in compliance with ethical guidelines approved by the Institutional Review Board (IRB). Informed consent will be obtained from participants or legal guardians, ensuring they fully understand the purpose, procedures, and potential risks of the study. All personal data will be anonymized to protect privacy.

10. Measures for Protecting Participant Privacy All personal data will be kept confidential. Data will be anonymized and stored securely, with access limited to the principal investigator and co-investigators. Video data will be encrypted and shared only with collaborating institutions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥19 years)
* Hospitalized patients with a Functional Ambulatory Category (FAC) score of ≤ 3 and who are bedridden.

Exclusion Criteria:

* Patients with significant cognitive impairment that prevents them from operating the app.
* Patients with severe pain or limited range of motion preventing participation in physical activity.
* Patients with severe biomechanical instability.
* Patients with significant sensory impairments (e.g., visual or auditory) that would hinder participation in the rehabilitation program.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility | From enrollment to the end of treatment at 2 weeks
  Record patient adherence to the rehabilitation program by entering the percentage of actual exercise time performed relative to the total prescribed exercise time.

SECONDARY OUTCOMES:
Safety | From enrollment to the end of treatment at 2 weeks
  Monitoring the number of occurrences of adverse events such as pain, falls, dizziness, and any other negative reactions during the rehabilitation sessions.

OTHER OUTCOMES:
Medical Research Council Sum Score (MRC-SS) | From enrollment to the end of treatment at 2 weeks
  Summation score of muscle strength based on MRC scale. Unit of Measure: Sum score (0 to 60, where a higher score indicates better overall muscle strength.)
Functional Ambulatory Category (FAC) | From enrollment to the end of treatment at 2 weeks
  Measurement of the level of ambulation and assistance required. Unit of Measure: FAC score (0 to 5, where a higher score indicates greater walking independence.)
Hand Grip Strength Test | From enrollment to the end of treatment at 2 weeks
  Measurement of grip strength using a dynamometer. Unit of Measure: Force (kg) (A higher value indicates better grip strength.)
Knee Extensor Test | From enrollment to the end of treatment at 2 weeks
  Assessment of knee extensor strength using a dynamometer. Unit of Measure: Force (N or kg) (A higher value indicates stronger knee extensor muscles.)
10-meter Walk Test (10MWT) | From enrollment to the end of treatment at 2 weeks
  Assessment of walking speed and functional mobility over a 10-meter distance. Unit of Measure: Time (seconds) or speed (m/s) (For time: A lower value indicates faster walking ability. For speed: A higher value indicates better walking performance.)
Mini-Mental State Examination (MMSE) | From enrollment to the end of treatment at 2 weeks
  Cognitive function assessment using the MMSE tool. Unit of Measure: MMSE score (0 to 30, where a higher score indicates better cognitive function.)
Satisfaction | From enrollment to the end of treatment at 2 weeks
  Assessment of patient satisfaction with the MORA app and its use during rehabilitation exercises.
  Measurement Tool: Overall satisfaction, interest about health, Application-related questions, exercise intensity questionnaire (5-point Likert scale) Unit of Measure: Satisfaction score (1 to 5, where a higher score indicates greater satisfaction.)
EQ-5D Health-Related Quality of Life | From enrollment to the end of treatment at 2 weeks
  Assessment of patient-reported quality of life using the EQ-5D questionnaire, covering mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Unit of Measure: Utility score (0 to 1) and VAS score (0 to 100)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Songpa-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
All individual patient data (IPD) used in this study will be handled in compliance with domestic privacy protection laws and relevant regulations. The privacy of study participants will be strictly safeguarded, and their personal information will not be used for purposes other than the study. When sharing data, only de-identified data that has been approved by the researchers after adequate request will be provided, and privacy protection and security will be prioritized throughout the process.